CLINICAL TRIAL: NCT03371355
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Dose Finding Study of ISIS 703802 (AKCEA-ANGPTL3-LRx) Administered Subcutaneously to Subjects With Hypertriglyceridemia, Type 2 Diabetes Mellitus (T2DM), and Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Study of ISIS 703802 in Participants With Hypertriglyceridemia, Type 2 Diabetes Mellitus, and Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Collaborators: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISIS 703802-CS2
Record Dates: First submitted 2017-11-27; First posted 2017-12-13 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2020-12

CONDITIONS: NAFLD; Diabetes Mellitus, Type 2; Hypertriglyceridemia; Fatty Liver, Nonalcoholic
Keywords: Type 2 Diabetes; Hepatic Steatosis; Triglycerides; AKCEA-ANGPTL3-Lrx; IONIS-ANGPTL3-Lrx; Fatty Liver; Fatty Liver Without Mention of Alcohol; Liver Fat; Liver Diseases; Diabetes Mellitus Type 2 in Nonobese; Diabetes Mellitus; Triglycerides High; High Triglycerides; Metabolic Disease; Endocrine System Diseases; Digestive System Disease; Glucose Metabolism Disorders; Vupanorsen
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Hypertriglyceridemia; Fatty Liver; Liver Diseases; Diabetes Mellitus; Metabolic Diseases; Endocrine System Diseases; Digestive System Diseases; Glucose Metabolism Disorders | interventions — IONIS-ANGPTL3-LRx; vupanorsen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pooled Placebo (Placebo Comparator): Participants from each cohort received placebo at a dose-matched volume of study drug, subcutaneously (SC).
  Interventions: Drug: Placebo
- Cohort B: ISIS 703802, 40 mg Q4W (Experimental): Participants received ISIS 703802, 40 milligrams (mg) SC once every 4 weeks for 6 doses.
  Interventions: Drug: ISIS 703802 40 mg
- Cohort C: ISIS 703802, 80 mg Q4W (Experimental): Participants received ISIS 703802, 80 mg SC once every 4 weeks for 6 doses.
  Interventions: Drug: ISIS 703802 80 mg
- Cohort A: ISIS 703802, 20 mg QW (Experimental): Participants received ISIS 703802, 20 mg once every week for 26 doses.
  Interventions: Drug: ISIS 703802 20 mg

INTERVENTIONS:
Drug: Placebo — Placebo (Matched with ISIS 703802)
  Other Names: Sterile Normal Saline (0.9% NaCl)
  Arms: Pooled Placebo
Drug: ISIS 703802 40 mg — ISIS 703802 40 mg, administered via SC injection, once every 4 weeks for 6 doses.
  Other Names: AKCEA-ANGPTL3-LRx; IONIS-ANGPTL3-LRx; Vupanorsen
  Arms: Cohort B: ISIS 703802, 40 mg Q4W
Drug: ISIS 703802 80 mg — ISIS 703802 80 mg, administered via SC injection, once every 4 weeks for 6 doses.
  Other Names: AKCEA-ANGPTL3-LRx; IONIS-ANGPTL3-LRx; Vupanorsen
  Arms: Cohort C: ISIS 703802, 80 mg Q4W
Drug: ISIS 703802 20 mg — ISIS 703802 20 mg, administered via SC injection, once every week for 26 doses.
  Other Names: AKCEA-ANGPTL3-LRx; IONIS-ANGPTL3-LRx; Vupanorsen
  Arms: Cohort A: ISIS 703802, 20 mg QW

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the safety, including tolerability, of ISIS 703802 and to assess the efficacy of different doses and dosing regimens of ISIS 703802 on glucose and lipid metabolism, and liver fat in participants with hypertriglyceridemia, Type 2 diabetes mellitus (T2DM), and nonalcoholic fatty liver disease (NAFLD).

ELIGIBILITY:
Key Inclusion Criteria:

* Plasma triglycerides (TG) at Screening greater than (>)150 milligrams per deciliter (mg/dL) and at qualification of >150 mg/dL.
* Documented history of hepatic steatosis with baseline magnetic resonance imaging (MRI) indicating hepatic fat fraction (HFF) greater than (>) 8%.
* Diagnosis of Type 2 diabetes mellitus with hemoglobin A1c (HbA1c) >6.5 and less than or equal to (≤) 10% at Screening.
* Must have been on a stable dose of oral antidiabetic therapy for a minimum of 3 months prior to Screening.
* Body mass index between 27- 40 kilograms per meter square (kg/m^2), inclusive, at Screening.

Key Exclusion Criteria:

* Type 1 diabetes mellitus.
* Active chronic liver disease, alcoholic liver disease, Wilson's disease hemochromatosis, primary biliary cirrhosis, primary sclerosing cholangitis, genetic hemochromatosis, known or suspected hepatocellular carcinoma, history of or planned liver transplant for end-stage liver disease of any etiology.
* Documented history of advanced liver fibrosis.
* History of cirrhosis and/or hepatic decompensation including ascites, hepatic encephalopathy, or variceal bleeding.
* History of clinically significant acute cardiac event within 6 months before Screening.
* History of heart failure with New York Heart Association (NYHA) greater than Class II.
* Use of Insulin or insulin analogs, glucagon-like peptide-1 (GLP-1) agonists, and peroxisome proliferator-activated receptor gamma (PPARᵞ) agonists (pioglitazone or rosiglitazone).
* Weight change >5% within 3 months before Screening.
* Conditions contraindicated for magnetic resonance imaging (MRI) procedures including any metal implant (example, heart pacemaker, rods, screws, aneurysm clips).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2020-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (37):
- United States (33):
  - Clinical Sites, Chandler, Arizona
  - Clinical Site, Fountain Hills, Arizona
  - Clinical Site, Glendale, Arizona
  - Clinical Site, Mesa, Arizona
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Huntington Park, California
  - Clinical Site, Los Angeles, California
  - Clinical Site, Montclair, California
  - Clinical Site, Panorama City, California
  - Clinical Site, Poway, California
  - Clinical Site, Boca Raton, Florida
  - Clinical Site, Jensen Beach, Florida
  - Clinical Site, Jupiter, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Port Saint Lucie, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Indianapolis, Indiana
  - Clinical Site, Louisville, Kentucky
  - Clinical Site, Edina, Minnesota
  - Clinical Site, Bridgeton, New Jersey
  - Clinical Site, Princeton, New Jersey
  - Clinical Site, Greensboro, North Carolina
  - Clinical Site, High Point, North Carolina
  - Clinical Site, Cincinnati, Ohio
  - Clinical Site, Charleston, South Carolina
  - Clinical Site, Austin, Texas
  - Clinical Site, Carrollton, Texas
  - Clinical Site, Dallas, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, Hurst, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical Site, Layton, Utah
- Canada (4):
  - Clinical Site, Hamilton, Ontario
  - Clinical Site, Toronto, Ontario
  - Clinical Site, Chicoutimi, Quebec
  - Clinical Site, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 42 study centers; 38 sites in the US and 4 sites in Canada.
Pre-assignment Details: A total of 525 participants were screened. 105 were randomized in a 1:1:1 ratio to Cohorts A, B, or C. In each cohort, participants were randomized in a 3:1 ratio to receive ISIS 703802 or matching volume of placebo.
Groups:
- Cohort A: ISIS 703802, 20 mg QW: Participants received ISIS 703802, 20 mg SC once every week for 26 doses.
Period: Overall Study
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Started | 27 | 26 | 26 | 26
Completed (Completed here refers to participants who completed study treatment.) | 26 | 24 | 22 | 19
Not Completed | 1 | 2 | 4 | 7
Not completed — Investigator judgment | 0 | 0 | 1 | 1
Not completed — Voluntary withdrawal | 1 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 2 | 3
Not completed — Reason not Specified | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Pooled Placebo: Participants from each cohort received placebo at a dose-matched volume of study drug, SC.
- Cohort B: ISIS 703802, 40 mg Q4W: Participants received ISIS 703802, 40 mg SC once every 4 weeks for 6 doses.
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW | Total
Number analyzed (Participants) | 27 | 26 | 26 | 26 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (7.29) | 52.0 (10.34) | 54.8 (6.04) | 56.0 (8.45) | 53.5 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 13 | 11 | 49
  Male | 11 | 17 | 13 | 15 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 13 | 11 | 17 | 65
  Not Hispanic or Latino | 3 | 13 | 15 | 9 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 1 | 5
  White | 25 | 23 | 24 | 25 | 97
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Fasting Triglycerides (TG) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 275.5 (110.38) | 414.9 (456.86) | 292.2 (130.98) | 311.8 (155.92) | 323.1 (257.20)
Angiopoietin Like 3 (ANGPTL3) [Mean (Standard Deviation); unit: micrograms per liter (μg/L)] | 114.85 (32.066) | 102.36 (28.923) | 111.86 (37.463) | 108.60 (42.722) | 109.47 (35.441)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 202.1 (43.64) | 200.7 (45.27) | 191.2 (61.63) | 182.4 (47.06) | 194.2 (49.78)
Non- High density lipoprotein cholesterol (Non-HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 162.7 (39.90) | 164.3 (47.50) | 154.1 (58.28) | 146.8 (46.79) | 157.0 (48.30)
High density lipoprotein cholesterol (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 39.4 (10.43) | 36.3 (10.54) | 37.1 (10.37) | 35.6 (9.89) | 37.1 (10.26)
Low Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] — LDL-C was calculated by using the precipitation method. Population: Number analyzed signifies the number of participants with data available for LDL-C.
  mg/dL
    number analyzed (Participants) | 25 | 23 | 23 | 25 | 96
    (all) | 111.5 (43.06) | 98.2 (36.13) | 101.0 (53.13) | 88.6 (37.69) | 99.8 (43.05)
Very Low Density Lipoprotein Cholesterol (VLDL-C) [Mean (Standard Deviation); unit: mg/dL] — Population: Number analyzed signifies the number of participants with data available for VLDL-C.
  mg/dL
    number analyzed (Participants) | 25 | 23 | 23 | 25 | 96
    (all) | 47.8 (12.90) | 52.6 (14.59) | 47.6 (9.92) | 49.6 (13.11) | 49.4 (12.71)
Apolipoprotein CIII (ApoCIII) [Mean (Standard Deviation); unit: mg/dL] | 14.48 (3.981) | 18.71 (11.024) | 15.54 (4.969) | 16.19 (5.562) | 16.21 (7.000)
Apolipoprotein A1 (ApoA1) [Mean (Standard Deviation); unit: mg/dL] | 141.3 (19.30) | 137.9 (21.12) | 139.1 (24.12) | 133.3 (20.18) | 137.9 (21.13)
Apolipoprotein B (ApoB) [Mean (Standard Deviation); unit: mg/dL] | 108.68 (25.254) | 105.90 (25.868) | 105.34 (36.160) | 95.48 (26.210) | 103.90 (28.721)
Apolipoprotein B48 (ApoB-48) [Mean (Standard Deviation); unit: mg/dL] | 2.63 (1.455) | 3.21 (2.239) | 3.20 (2.863) | 3.48 (3.228) | 3.13 (2.511)
Apolipoprotein B100 (ApoB-100) [Mean (Standard Deviation); unit: mg/dL] | 105.89 (25.699) | 102.48 (25.740) | 102.14 (35.392) | 91.79 (25.871) | 100.62 (28.540)
Lipoprotein-a (Lp[a]) [Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)] | 51.7 (66.79) | 58.2 (74.74) | 46.7 (74.88) | 38.3 (54.81) | 48.8 (67.69)
Free Fatty Acid (FFA) [Mean (Standard Deviation); unit: millimole per liter (mmol/L)] | 0.62 (0.261) | 0.66 (0.266) | 0.61 (0.237) | 0.58 (0.213) | 0.62 (0.243)
Insulin [Mean (Standard Deviation); unit: milli international units per liter] — Population: Number analyzed signifies the number of participants with data available for insulin.
  milli international units per liter
    number analyzed (Participants) | 27 | 26 | 25 | 25 | 103
    (all) | 26.35 (16.965) | 21.35 (12.602) | 26.32 (15.353) | 23.19 (12.887) | 24.31 (14.542)
Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] — Population: Number analyzed signifies the number of participants with data available for plasma glucose.
  mg/dL
    number analyzed (Participants) | 27 | 26 | 25 | 25 | 103
    (all) | 188.6 (59.06) | 182.6 (58.87) | 201.4 (52.16) | 164.6 (47.69) | 184.4 (55.55)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: index] — HOMA-IR is a method used to quantify insulin resistance. HOMA-IR is expressed as the following: HOMA-IR = fasting serum insulin (microunits per milliliter [μU/Ml]) * fasting plasma glucose (millimoles/liter [mmol/L])/22.5. Population: Number analyzed signifies the number of participants with data available for HOMA-IR.
  index
    number analyzed (Participants) | 27 | 26 | 25 | 25 | 103
    (all) | 12.40 (8.548) | 9.42 (6.178) | 13.02 (8.331) | 9.54 (6.278) | 11.10 (7.500)
Fructosamine [Mean (Standard Deviation); unit: micromoles per liter (μmol/L)] | 325.2 (49.62) | 302.7 (65.51) | 317.6 (59.33) | 312.9 (48.19) | 314.7 (55.85)
Glycated Albumin [Mean (Standard Deviation); unit: grams per deciliter (g/dL)] | 0.84 (0.183) | 0.74 (0.254) | 0.80 (0.216) | 0.79 (0.187) | 0.79 (0.211)
Hemoglobin A1C (HbA1C) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.30 (1.260) | 8.04 (1.113) | 8.36 (1.091) | 8.19 (0.901) | 8.22 (1.091)
Hepatic Fat Fraction (HFF) [Mean (Standard Deviation); unit: percentage (Hepatic Fat Fraction)] | 16.84 (6.144) | 17.17 (6.150) | 17.23 (7.262) | 19.32 (10.445) | 17.63 (7.642)
Subcutaneous Adipose Tissue (SAT) [Mean (Standard Deviation); unit: millimeters square (mm^2)] | 2634.49 (1235.433) | 3076.36 (1114.681) | 3021.37 (1080.432) | 2701.94 (1000.756) | 2856.41 (1113.220)
Visceral Adipose Tissue (VAT), [Mean (Standard Deviation); unit: mm^2] | 2275.05 (605.492) | 2690.34 (888.431) | 2826.84 (1105.086) | 2773.11 (894.630) | 2637.85 (903.168)
Fatty Liver Index (FLI) [Mean (Standard Deviation); unit: index] — The FLI was calculated by the following formula: FLI =(e0.953×loge[triglycerides]+0.139× Body Mass Index[BMI]+0.718×loge Gamma- Glutamyl Transferase [GGT]+0.053×waistcircumference-15.745)/ (1 +e0.953×loge[triglycerides]+0.139×BMI+0.718×loge [GGT]+0.053×waistcircumference-15.745) × 100. Population: Number analyzed signifies the number of participants with data available for FLI.
  index
    number analyzed (Participants) | 27 | 25 | 26 | 26 | 104
    (all) | 77.20 (22.618) | 85.55 (12.802) | 83.16 (19.846) | 84.45 (13.926) | 82.51 (17.907)
Body Weight [Mean (Standard Deviation); unit: kg] | 79.3 (10.64) | 92.5 (16.66) | 90.7 (20.83) | 92.0 (16.39) | 88.5 (17.15)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] | 30.3 (3.03) | 32.8 (3.97) | 32.1 (3.84) | 32.3 (4.19) | 31.9 (3.84)
Waist to Hip Ratio [Mean (Standard Deviation); unit: ratio] — Population: Number analyzed signifies the number of participants with data available for waist to hip ratio.
  ratio
    number analyzed (Participants) | 27 | 26 | 25 | 26 | 104
    (all) | 0.98 (0.070) | 1.05 (0.225) | 1.01 (0.216) | 0.97 (0.068) | 1.00 (0.163)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Fasting Triglycerides Level at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the log ratio of Primary Analysis Time Point to Baseline. The estimate of the log ratio was converted back to the original scale and percent change was calculated using formula: = (ratio of Primary Analysis Time Point to Baseline - 1) × 100.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 27 | 26 | 26 | 26
percent change | -16 [-29 to 0] | -36 [-47 to -23] | -53 [-60 to -43] | -47 [-57 to -35]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.0343, ANCOVA; Mean Difference in % CFB = -24, 95% CI 2-sided [-41 to -2] — Mean difference in percent (%) change from baseline (CFB) based on difference in least square mean (LSM) of log (Primary Analysis Time Point/Baseline) was estimated
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -44, 95% CI 2-sided [-56 to -28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.0009, ANCOVA; Mean Difference in % CFB = -37, 95% CI 2-sided [-52 to -17] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Angiopoietin-Like 3 Protein at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug. Here, overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/L
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 23 | 17
μg/L | 6.77 [-2.09 to 15.62] | -43.11 [-52.27 to -33.94] | -64.89 [-74.26 to -55.53] | -52.98 [-63.99 to -41.96]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -49.87, 95% CI 2-sided [-62.68 to -37.06]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -71.66, 95% CI 2-sided [-84.47 to -58.85]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -59.74, 95% CI 2-sided [-74.04 to -45.44]

3. Secondary Outcome: Change From Baseline in TC, LDL-C, HDL-C, VLDL-C, Non-HDL-C, ApoB (ApoB-48, ApoB-100), ApoCIII, and ApoAI at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug. Here, 'number analyzed' (n) signifies participants evaluable for this outcome measure for each specified category.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 27 | 26 | 26 | 26
mg/dL
  TC: number analyzed (Participants) | 26 | 23 | 23 | 17
  TC | -4.8 [-15.19 to 5.51] | -21.3 [-32.35 to -10.31] | -41.9 [-52.88 to -30.89] | -36.5 [-49.38 to -23.58]
  LDL-C: number analyzed (Participants) | 23 | 19 | 23 | 17
  LDL-C | -2.5 [-11.21 to 6.14] | 5.0 [-4.78 to 14.70] | -11.1 [-20.38 to -1.90] | -11.3 [-21.76 to -0.84]
  HDL-C: number analyzed (Participants) | 26 | 23 | 23 | 17
  HDL-C | 2.2 [-0.38 to 4.69] | -0.6 [-3.25 to 2.14] | -6.4 [-9.13 to -3.77] | -2.0 [-5.11 to 1.12]
  VLDL-C: number analyzed (Participants) | 23 | 19 | 23 | 17
  VLDL-C | -6.5 [-11.64 to -1.34] | -15.6 [-21.47 to -9.78] | -21.9 [-27.41 to -16.36] | -17.3 [-23.48 to -11.13]
  Non-HDL-C: number analyzed (Participants) | 26 | 23 | 23 | 17
  Non-HDL-C | -7.0 [-17.45 to 3.44] | -20.9 [-32.01 to -9.70] | -35.4 [-46.54 to -24.33] | -34.4 [-47.39 to -21.34]
  ApoB: number analyzed (Participants) | 26 | 23 | 23 | 17
  ApoB | -3.63 [-9.98 to 2.71] | -6.08 [-12.82 to 0.66] | -13.46 [-20.20 to -6.72] | -8.91 [-16.91 to -0.91]
  ApoB: ApoB-48: number analyzed (Participants) | 26 | 24 | 23 | 17
  ApoB: ApoB-48 | -0.139 [-0.90 to 0.62] | -1.140 [-1.93 to -0.35] | -1.942 [-2.75 to -1.14] | -1.230 [-2.16 to -0.30]
  ApoB: ApoB-100: number analyzed (Participants) | 26 | 23 | 23 | 17
  ApoB: ApoB-100 | -3.757 [-9.94 to 2.43] | -4.643 [-11.21 to 1.92] | -11.346 [-17.91 to -4.78] | -7.174 [-14.97 to 0.62]
  ApoCIII: number analyzed (Participants) | 26 | 24 | 23 | 17
  ApoCIII | -0.729 [-2.58 to 1.12] | -5.482 [-7.42 to -3.54] | -9.228 [-11.18 to -7.28] | -7.588 [-9.86 to -5.32]
  ApoA1: number analyzed (Participants) | 26 | 23 | 23 | 17
  ApoA1 | 5.0 [-1.11 to 11.15] | -11.8 [-18.32 to -5.30] | -30.1 [-36.63 to -23.65] | -16.1 [-23.68 to -8.57]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; TC; Test type: Superiority; p = 0.0327, ANCOVA; Least Squares Mean Difference = -16.5, 95% CI 2-sided [-31.59 to -1.39]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; TC; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -37.0, 95% CI 2-sided [-52.15 to -21.94]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; TC; Test type: Superiority; p = 0.0003, ANCOVA; Least Squares Mean Difference = -31.6, 95% CI 2-sided [-48.23 to -15.05]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; LDL-C; Test type: Superiority; p = 0.2560, ANCOVA; Least Squares Mean Difference = 7.5, 95% CI 2-sided [-5.55 to 20.54]
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; LDL-C; Test type: Superiority; p = 0.1795, ANCOVA; Least Squares Mean Difference = -8.6, 95% CI 2-sided [-21.26 to 4.05]
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; LDL-C; Test type: Superiority; p = 0.2065, ANCOVA; Least Squares Mean Difference = -8.8, 95% CI 2-sided [-22.48 to 4.95]
Statistical Analysis 7: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; HDL-C; Test type: Superiority; p = 0.1515, ANCOVA; Least Squares Mean Difference = -2.7, 95% CI 2-sided [-6.43 to 1.01]
Statistical Analysis 8: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; HDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -8.6, 95% CI 2-sided [-12.29 to -4.91]
Statistical Analysis 9: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; HDL-C; Test type: Superiority; p = 0.0436, ANCOVA; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-8.18 to -0.12]
Statistical Analysis 10: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; VLDL-C; Test type: Superiority; p = 0.0224, ANCOVA; Least Squares Mean Difference = -9.1, 95% CI 2-sided [-16.94 to -1.33]
Statistical Analysis 11: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; VLDL-C; Test type: Superiority; p = 0.0001, ANCOVA; Least Squares Mean Difference = -15.4, 95% CI 2-sided [-22.94 to -7.84]
Statistical Analysis 12: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; VLDL-C; Test type: Superiority; p = 0.0091, ANCOVA; Least Squares Mean Difference = -10.8, 95% CI 2-sided [-18.86 to -2.78]
Statistical Analysis 13: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Non-HDL-C; Test type: Superiority; p = 0.0748, ANCOVA; Least Squares Mean Difference = -13.9, 95% CI 2-sided [-29.12 to 1.42]
Statistical Analysis 14: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Non-HDL-C; Test type: Superiority; p = 0.0004, ANCOVA; Least Squares Mean Difference = -28.4, 95% CI 2-sided [-43.68 to -13.18]
Statistical Analysis 15: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Non-HDL-C; Test type: Superiority; p = 0.0016, ANCOVA; Least Squares Mean Difference = -27.4, 95% CI 2-sided [-44.08 to -10.64]
Statistical Analysis 16: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoB; Test type: Superiority; p = 0.6005, ANCOVA; Least Squares Mean Difference = -2.44, 95% CI 2-sided [-11.68 to 6.80]
Statistical Analysis 17: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoB; Test type: Superiority; p = 0.0374, ANCOVA; Least Squares Mean Difference = -9.83, 95% CI 2-sided [-19.07 to -0.59]
Statistical Analysis 18: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoB; Test type: Superiority; p = 0.3100, ANCOVA; Least Squares Mean Difference = -5.28, 95% CI 2-sided [-15.55 to 5.00]
Statistical Analysis 19: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoB-48; Test type: Superiority; p = 0.0728, ANCOVA; Least Squares Mean Difference = -1.002, 95% CI 2-sided [-2.10 to 0.09]
Statistical Analysis 20: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoB-48; Test type: Superiority; p = 0.0018, ANCOVA; Least Squares Mean Difference = -1.803, 95% CI 2-sided [-2.91 to -0.69]
Statistical Analysis 21: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoB-48; Test type: Superiority; p = 0.0759, ANCOVA; Least Squares Mean Difference = -1.091, 95% CI 2-sided [-2.30 to 0.12]
Statistical Analysis 22: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoB-100; Test type: Superiority; p = 0.8451, ANCOVA; Least Squares Mean Difference = -0.887, 95% CI 2-sided [-9.89 to 8.11]
Statistical Analysis 23: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoB-100; Test type: Superiority; p = 0.0973, ANCOVA; Least Squares Mean Difference = -7.590, 95% CI 2-sided [-16.59 to 1.41]
Statistical Analysis 24: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoB-100; Test type: Superiority; p = 0.5000, ANCOVA; Least Squares Mean Difference = -3.418, 95% CI 2-sided [-13.45 to 6.61]
Statistical Analysis 25: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoCIII; Test type: Superiority; p = 0.0008, ANCOVA; Least Squares Mean Difference = -4.753, 95% CI 2-sided [-7.47 to -2.03]
Statistical Analysis 26: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoCIII; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -8.499, 95% CI 2-sided [-11.18 to -5.82]
Statistical Analysis 27: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoCIII; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -6.860, 95% CI 2-sided [-9.78 to -3.93]
Statistical Analysis 28: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoA1; Test type: Superiority; p = 0.0003, ANCOVA; Least Squares Mean Difference = -16.8, 95% CI 2-sided [-25.80 to -7.85]
Statistical Analysis 29: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoA1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -35.2, 95% CI 2-sided [-44.07 to -26.24]
Statistical Analysis 30: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoA1; Test type: Superiority; p < 0.0001, ANCOVA; Least Squares Mean Difference = -21.1, 95% CI 2-sided [-30.89 to -11.39]

4. Secondary Outcome: Change From Baseline in Free Fatty Acid (FFA) at Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 23 | 17
mmol/L | -0.0734 [-0.15 to 0.01] | -0.0607 [-0.15 to 0.02] | -0.0878 [-0.17 to 0.00] | -0.0881 [-0.19 to 0.01]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.8299, ANCOVA; Least Squares Mean Difference = 0.0128, 95% CI 2-sided [-0.10 to 0.13]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.8102, ANCOVA; Least Squares Mean Difference = -0.0144, 95% CI 2-sided [-0.13 to 0.10]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.8223, ANCOVA; Least Squares Mean Difference = -0.0146, 95% CI 2-sided [-0.14 to 0.11]

5. Secondary Outcome: Change From Baseline in Lipoprotein(a) (Lp[a]) at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 23 | 23 | 17
nmol/L | -1.1 [-6.67 to 4.51] | 6.8 [0.76 to 12.75] | 0.5 [-5.47 to 6.44] | -2.8 [-9.74 to 4.15]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Lp(a); Test type: Superiority; p = 0.0604, ANCOVA; Least Squares Mean Difference = 7.8, 95% CI 2-sided [-0.35 to 16.02]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Lp(a); Test type: Superiority; p = 0.7048, ANCOVA; Least Squares Mean Difference = 1.6, 95% CI 2-sided [-6.61 to 9.74]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Lp(a); Test type: Superiority; p = 0.7024, ANCOVA; Least Squares Mean Difference = -1.7, 95% CI 2-sided [-10.65 to 7.20]

6. Secondary Outcome: Percent Change From Baseline in ANGPTL3, TC, LDL-C, HDL-C, VLDL-C, Non-HDL-C, ApoB (ApoB-48, ApoB-100), ApoCIII, ApoAI, FFA, and Lp(a) at Primary Analysis Time Point
Description: as for outcome 1
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug. Here, 'n' signifies participants evaluable for this outcome measure for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 27 | 26 | 26 | 26
percent change
  ANGPTL3: number analyzed (Participants) | 26 | 24 | 23 | 17
  ANGPTL3 | 8 [-6 to 23] | -41 [-48 to -32] | -59 [-64 to -53] | -54 [-61 to -46]
  TC: number analyzed (Participants) | 26 | 23 | 23 | 17
  TC | -2 [-8 to 4] | -11 [-16 to -5] | -21 [-26 to -16] | -19 [-25 to -13]
  LDL-C: number analyzed (Participants) | 23 | 19 | 23 | 17
  LDL-C | 0 [-8 to 9] | 6 [-4 to 17] | -7 [-15 to 2] | -12 [-21 to -3]
  HDL-C: number analyzed (Participants) | 26 | 23 | 23 | 17
  HDL-C | 7 [-2 to 16] | -2 [-10 to 8] | -18 [-25 to -11] | -4 [-13 to 6]
  VLDL-C: number analyzed (Participants) | 23 | 19 | 23 | 17
  VLDL-C | -14 [-26 to 0] | -35 [-45 to -23] | -47 [-55 to -37] | -40 [-50 to -28]
  Non-HDL-C: number analyzed (Participants) | 26 | 23 | 23 | 17
  Non-HDL-C | -4 [-11 to 3] | -13 [-20 to -7] | -21 [-27 to -15] | -22 [-29 to -15]
  ApoB: number analyzed (Participants) | 26 | 23 | 23 | 17
  ApoB | -3 [-9 to 3] | -7 [-12 to 0] | -12 [-17 to -6] | -10 [-17 to -3]
  ApoB: ApoB-48: number analyzed (Participants) | 26 | 24 | 23 | 17
  ApoB: ApoB-48 | -21 [-40 to 5] | -44 [-58 to -25] | -62 [-72 to -49] | -38 [-56 to -12]
  ApoB: ApoB-100: number analyzed (Participants) | 26 | 23 | 23 | 17
  ApoB: ApoB-100 | -3 [-9 to 3] | -5 [-11 to 1] | -10 [-16 to -4] | -9 [-15 to -1]
  ApoCIII: number analyzed (Participants) | 26 | 24 | 23 | 17
  ApoCIII | -6 [-22 to 14] | -40 [-51 to -27] | -61 [-68 to -52] | -50 [-61 to -37]
  ApoA1: number analyzed (Participants) | 26 | 23 | 23 | 17
  ApoA1 | 3 [-4 to 11] | -9 [-15 to -2] | -24 [-29 to -18] | -12 [-19 to -4]
  FFA: number analyzed (Participants) | 26 | 24 | 23 | 17
  FFA | -11 [-24 to 4] | -12 [-25 to 3] | -18 [-31 to -4] | -11 [-27 to 8]
  Lp(a): number analyzed (Participants) | 26 | 23 | 23 | 17
  Lp(a) | 3 [-8 to 15] | -4 [-15 to 8] | -3 [-14 to 9] | -1 [-14 to 13]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ANGPTL3; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -45, 95% CI 2-sided [-54 to -33] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ANGPTL3; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -62, 95% CI 2-sided [-69 to -54] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ANGPTL3; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -58, 95% CI 2-sided [-66 to -47] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; TC; Test type: Superiority; p = 0.0309, ANCOVA; Mean Difference in % CFB = -9, 95% CI 2-sided [-16 to -1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; TC; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -19, 95% CI 2-sided [-26 to -12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; TC; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -17, 95% CI 2-sided [-25 to -9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; LDL-C; Test type: Superiority; p = 0.4016, ANCOVA; Mean Difference in % CFB = 6, 95% CI 2-sided [-7 to 21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; LDL-C; Test type: Superiority; p = 0.2589, ANCOVA; Mean Difference in % CFB = -7, 95% CI 2-sided [-18 to 6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; LDL-C; Test type: Superiority; p = 0.0616, ANCOVA; Mean Difference in % CFB = -12, 95% CI 2-sided [-24 to 1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; HDL-C; Test type: Superiority; p = 0.1918, ANCOVA; Mean Difference in % CFB = -8, 95% CI 2-sided [-18 to 4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; HDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -24, 95% CI 2-sided [-32 to -14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; HDL-C; Test type: Superiority; p = 0.1132, ANCOVA; Mean Difference in % CFB = -10, 95% CI 2-sided [-21 to 3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; VLDL-C; Test type: Superiority; p = 0.0177, ANCOVA; Mean Difference in % CFB = -24, 95% CI 2-sided [-40 to -5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; VLDL-C; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -38, 95% CI 2-sided [-51 to -23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; VLDL-C; Test type: Superiority; p = 0.0033, ANCOVA; Mean Difference in % CFB = -30, 95% CI 2-sided [-45 to -12] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Non-HDL-C; Test type: Superiority; p = 0.0523, ANCOVA; Mean Difference in % CFB = -10, 95% CI 2-sided [-18 to 0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Non-HDL-C; Test type: Superiority; p = 0.0002, ANCOVA; Mean Difference in % CFB = -18, 95% CI 2-sided [-26 to -9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Non-HDL-C; Test type: Superiority; p = 0.0004, ANCOVA; Mean Difference in % CFB = -19, 95% CI 2-sided [-28 to -9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoB; Test type: Superiority; p = 0.4204, ANCOVA; Mean Difference in % CFB = -3, 95% CI 2-sided [-12 to 5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoB; Test type: Superiority; p = 0.0441, ANCOVA; Mean Difference in % CFB = -9, 95% CI 2-sided [-16 to 0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoB; Test type: Superiority; p = 0.1324, ANCOVA; Mean Difference in % CFB = -7, 95% CI 2-sided [-16 to 2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoB-48; Test type: Superiority; p = 0.1009, ANCOVA; Mean Difference in % CFB = -29, 95% CI 2-sided [-53 to 7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoB-48; Test type: Superiority; p = 0.0005, ANCOVA; Mean Difference in % CFB = -52, 95% CI 2-sided [-68 to -28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoB-48; Test type: Superiority; p = 0.3004, ANCOVA; Mean Difference in % CFB = -21, 95% CI 2-sided [-50 to 24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 25: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoB-100; Test type: Superiority; p = 0.6135, ANCOVA; Mean Difference in % CFB = -2, 95% CI 2-sided [-10 to 7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 26: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoB-100; Test type: Superiority; p = 0.1127, ANCOVA; Mean Difference in % CFB = -7, 95% CI 2-sided [-15 to 2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 27: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoB-100; Test type: Superiority; p = 0.2576, ANCOVA; Mean Difference in % CFB = -5, 95% CI 2-sided [-14 to 4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 28: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoCIII; Test type: Superiority; p = 0.0017, ANCOVA; Mean Difference in % CFB = -36, 95% CI 2-sided [-52 to -16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 29: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoCIII; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -58, 95% CI 2-sided [-68 to -45] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 30: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoCIII; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -47, 95% CI 2-sided [-61 to -29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 31: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ApoAI; Test type: Superiority; p = 0.0193, ANCOVA; Mean Difference in % CFB = -11, 95% CI 2-sided [-20 to -2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 32: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ApoAI; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference in % CFB = -26, 95% CI 2-sided [-33 to -19] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 33: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ApoAI; Test type: Superiority; p = 0.0063, ANCOVA; Mean Difference in % CFB = -14, 95% CI 2-sided [-23 to -4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 34: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; FFA; Test type: Superiority; p = 0.8873, ANCOVA; Mean Difference in % CFB = -2, 95% CI 2-sided [-21 to 23] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 35: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; FFA; Test type: Superiority; p = 0.4404, ANCOVA; Mean Difference in % CFB = -8, 95% CI 2-sided [-27 to 15] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 36: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; FFA; Test type: Superiority; p = 0.9665, ANCOVA; Mean Difference in % CFB] = -1, 95% CI 2-sided [-22 to 27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 37: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Lp[a]; Test type: Superiority; p = 0.4133, ANCOVA; Mean Difference in % CFB] = -7, 95% CI 2-sided [-21 to 10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 38: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Lp[a]; Test type: Superiority; p = 0.4750, ANCOVA; Mean Difference in % CFB] = -6, 95% CI 2-sided [-20 to 11] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 39: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Lp[a]; Test type: Superiority; p = 0.6354, ANCOVA; Mean Difference in % CFB] = -4, 95% CI 2-sided [-20 to 15] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 23 | 23 | 16
mg/dL | -4.4 [-21.74 to 12.95] | -21.6 [-40.05 to -3.17] | 9.4 [-9.53 to 28.40] | -2.2 [-25.33 to 20.90]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.1799, ANCOVA; Least Squares Mean Difference = -17.2, 95% CI 2-sided [-42.53 to 8.10]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.2867, ANCOVA; Least Squares Mean Difference = 13.8, 95% CI 2-sided [-11.83 to 39.49]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.8812, ANCOVA; Least Squares Mean Difference = 2.2, 95% CI 2-sided [-26.78 to 31.14]

8. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of HbA1c
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 24 | 22 | 19
percentage of HbA1c | 0.19 [-0.27 to 0.64] | -0.09 [-0.56 to 0.37] | 0.26 [-0.22 to 0.75] | 0.35 [-0.18 to 0.87]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.3995, ANCOVA; Least Squares Mean Difference = -0.28, 95% CI 2-sided [-0.94 to 0.38]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.8155, ANCOVA; Least Squares Mean Difference = 0.08, 95% CI 2-sided [-0.59 to 0.75]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.6466, ANCOVA; Least Squares Mean Difference = 0.16, 95% CI 2-sided [-0.54 to 0.86]

9. Secondary Outcome: Change From Baseline in Fasting Insulin at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: milli-international units per liter
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 23 | 23 | 16
milli-international units per liter | -0.10 [-5.74 to 5.55] | -1.48 [-7.51 to 4.54] | -0.23 [-6.37 to 5.91] | 3.48 [-3.94 to 10.9]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.7393, ANCOVA; Least Squares Mean Difference = 1.39, 95% CI 2-sided [-9.66 to 6.89]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.9744, ANCOVA; Least Squares Mean Difference = -0.13, 95% CI 2-sided [-8.45 to 8.18]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.4477, ANCOVA; Least Squares Mean Difference = 3.58, 95% CI 2-sided [-5.75 to 12.91]

10. Secondary Outcome: Change From Baseline in and HOMA-IR at the Primary Analysis Time Point
Description: HOMA-IR is a method used to quantify insulin resistance. HOMA-IR is expressed as the following: HOMA-IR = fasting serum insulin (μU/mL) * fasting plasma glucose (mmol/L)/22.5. A negative change from Baseline indicates improvement. An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 23 | 23 | 16
index | -0.119 [-3.47 to 3.24] | -1.914 [-5.50 to 1.67] | 0.141 [-3.52 to 3.80] | 2.013 [-2.41 to 6.44]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.4710, ANCOVA; Least Squares Mean Difference = -1.794, 95% CI 2-sided [-6.72 to 3.14]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.9169, ANCOVA; Least Squares Mean Difference = 0.260, 95% CI 2-sided [-4.68 to 5.20]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.4484, ANCOVA; Least Squares Mean Difference = 2.133, 95% CI 2-sided [-3.44 to 7.70]

11. Secondary Outcome: Change From Baseline in Fructosamine at Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 23 | 17
μmol/L | 13.2 [-5.40 to 31.80] | -10.0 [-29.34 to 9.40] | 1.8 [-17.92 to 21.44] | 15.1 [-7.74 to 38.04]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.0916, ANCOVA; Least Squares Mean Difference = -23.2, 95% CI 2-sided [-50.17 to 3.83]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.4032, ANCOVA; Least Squares Mean Difference = -11.4, 95% CI 2-sided [-38.51 to 15.63]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.8959, ANCOVA; Least Squares Mean Difference = 1.9, 95% CI 2-sided [-27.56 to 31.45]

12. Secondary Outcome: Change From Baseline in Glycated Albumin at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: grams per deciliter (g/dL)
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 23 | 17
grams per deciliter (g/dL) | -0.0033 [-0.07 to 0.07] | -0.0553 [-0.13 to 0.02] | -0.0133 [-0.09 to 0.06] | 0.0280 [-0.06 to 0.12]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.3202, ANCOVA; Least Squares Mean Difference = -0.0520, 95% CI 2-sided [-0.16 to 0.05]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.8485, ANCOVA; Least Squares Mean Difference = -0.0100, 95% CI 2-sided [-0.11 to 0.09]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.5812, ANCOVA; Least Squares Mean Difference = 0.0314, 95% CI 2-sided [-0.08 to 0.14]

13. Secondary Outcome: Change From Baseline in Weight at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 25 | 22
kg | -1.00 [-2.19 to 0.18] | -0.57 [-1.76 to 0.62] | -0.99 [-2.15 to 0.17] | -1.33 [-2.57 to -0.09]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.6157, ANCOVA; Least Squares Mean Difference = 0.43, 95% CI 2-sided [-1.28 to 2.15]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.9869, ANCOVA; Least Squares Mean Difference = 0.01, 95% CI 2-sided [-1.66 to 1.69]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.7084, ANCOVA; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-2.07 to 1.42]

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 25 | 22
millimeters of mercury (mmHg)
  SBP | -1.66 [-6.66 to 3.33] | 1.13 [-4.07 to 6.34] | 0.42 [-4.67 to 5.51] | -3.29 [-8.76 to 2.17]
  DBP | -2.35 [-5.71 to 1.00] | 1.75 [-1.70 to 5.20] | 1.13 [-2.26 to 4.52] | -0.73 [-4.35 to 2.88]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; SBP; Test type: Superiority; p = 0.4431, ANCOVA; Least Squares Mean Difference = 2.79, 95% CI 2-sided [-4.41 to 10.00]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; SBP; Test type: Superiority; p = 0.5630, ANCOVA; Least Squares Mean Difference = 2.08, 95% CI 2-sided [-5.05 to 9.22]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; SBP; Test type: Superiority; p = 0.6634, ANCOVA; Least Squares Mean Difference = -1.63, 95% CI 2-sided [-9.06 to 5.79]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; DBP; Test type: Superiority; p = 0.0937, ANCOVA; Least Squares Mean Difference = 4.11, 95% CI 2-sided [-0.71 to 8.92]
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; DBP; Test type: Superiority; p = 0.1522, ANCOVA; Least Squares Mean Difference = 3.49, 95% CI 2-sided [-1.31 to 8.28]
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; DBP; Test type: Superiority; p = 0.5188, ANCOVA; Least Squares Mean Difference = 1.62, 95% CI 2-sided [-3.35 to 6.59]

15. Secondary Outcome: Percent Change From Baseline in Weight, SBP and DBP at Primary Analysis Time Point
Description: An ANCOVA model was performed on the percent change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C6
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 25 | 22
percent change
  Weight | -0.98 [-2.23 to 0.27] | -0.40 [-1.66 to 0.85] | -1.10 [-2.32 to 0.12] | -1.38 [-2.69 to -0.07]
  SBP | -0.55 [-4.57 to 3.46] | 1.80 [-2.38 to 5.98] | 0.68 [-3.41 to 4.77] | -1.79 [-6.17 to 2.60]
  DBP | -1.83 [-6.22 to 2.56] | 3.18 [-1.33 to 7.69] | 2.11 [-2.32 to 6.54] | -0.13 [-4.85 to 4.60]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Weight; Test type: Superiority; p = 0.5299, ANCOVA; Least Squares Mean Difference = 0.57, 95% CI 2-sided [-1.24 to 2.39]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Weight; Test type: Superiority; p = 0.8919, ANCOVA; Least Squares Mean Difference = -0.12, 95% CI 2-sided [-1.89 to 1.65]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Weight; Test type: Superiority; p = 0.6653, ANCOVA; Least Squares Mean Difference = -0.40, 95% CI 2-sided [-2.25 to 1.44]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; SBP; Test type: Superiority; p = 0.4213, ANCOVA; Least Squares Mean Difference = 2.35, 95% CI 2-sided [-3.43 to 8.14]
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; SBP; Test type: Superiority; p = 0.6696, ANCOVA; Least Squares Mean Difference = 1.23, 95% CI 2-sided [-4.49 to 6.96]
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; SBP; Test type: Superiority; p = 0.6819, ANCOVA; Least Squares Mean Difference = -1.23, 95% CI 2-sided [-7.20 to 4.73]
Statistical Analysis 7: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; DBP; Test type: Superiority; p = 0.1171, ANCOVA; Least Squares Mean Difference = 5.01, 95% CI 2-sided [-1.28 to 11.31]
Statistical Analysis 8: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; DBP; Test type: Superiority; p = 0.2155, ANCOVA; Least Squares Mean Difference = 3.94, 95% CI 2-sided [-2.33 to 10.21]
Statistical Analysis 9: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; DBP; Test type: Superiority; p = 0.6034, ANCOVA; Least Squares Mean Difference = 1.70, 95% CI 2-sided [-4.79 to 8.20]

16. Secondary Outcome: Change From Baseline in Hepatic Fat Fraction (HFF) by Magnetic Resonance Imaging-Derived Proton Density Fat Fraction (MRI-PDFF) at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage (Hepatic Fat Fraction)
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 23 | 22 | 19
percentage (Hepatic Fat Fraction) | -1.69 [-4.09 to 0.71] | -0.71 [-3.21 to 1.78] | 2.39 [-0.16 to 4.94] | -0.12 [-2.87 to 2.64]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.5752, ANCOVA; Least Squares Mean Difference = 0.98, 95% CI 2-sided [-2.48 to 4.44]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.0230, ANCOVA; Least Squares Mean Difference = 4.09, 95% CI 2-sided [0.58 to 7.59]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.3965, ANCOVA; Least Squares Mean Difference = 1.57, 95% CI 2-sided [-2.10 to 5.25]

17. Secondary Outcome: Percent Change From Baseline in Hepatic Fat Fraction (HFF) by Magnetic Resonance Imaging-Derived Proton Density Fat Fraction (MRI-PDFF) at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the percent change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 23 | 22 | 19
percent change | -7.09 [-23.63 to 9.45] | 5.34 [-11.83 to 22.52] | 18.94 [1.38 to 36.51] | 5.18 [-13.80 to 24.15]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.3023, ANCOVA; Least Squares Mean Difference = 12.44, 95% CI 2-sided [-11.39 to 36.26]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.0350, ANCOVA; Least Squares Mean Difference = 26.03, 95% CI 2-sided [1.87 to 50.19]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.3374, ANCOVA; Least Squares Mean Difference = 12.27, 95% CI 2-sided [-13.02 to 37.55]

18. Secondary Outcome: Percentage of Participants With HFF ≤ 8% by MRI-PDFF at the Primary Analysis Time Point
Description: The percentage of participants who achieved HFF ≤ 8% at the Primary Analysis Time Point was compared between each ISIS 703802 treatment group and pooled placebo group using a logistic regression model.
Time Frame: Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 23 | 22 | 19
percentage of participants | 16.0 | 8.7 | 4.5 | 15.8

19. Secondary Outcome: Change From Baseline in Fatty Liver Index (FLI) at the Primary Analysis Time Point
Description: The FLI was calculated by the following formula: FLI =(e0.953×loge[triglycerides]+0.139× Body Mass Index [BMI]+0.718×loge Gamma- Glutamyl Transferase [GGT]+0.053×waistcircumference-15.745)/ (1 + e0.953×loge[triglycerides]+0.139×BMI+0.718×loge [GGT]+0.053×waistcircumference-15.745) × 100. An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: index
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 23 | 24 | 22
index | -3.50 [-8.21 to 1.22] | -6.08 [-11.08 to -1.09] | -9.21 [-13.99 to -4.44] | -8.07 [-13.06 to -3.07]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.4583, ANCOVA; Least Squares Mean Difference = -2.59, 95% CI 2-sided [-9.49 to 4.31]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.0943, ANCOVA; Least Squares Mean Difference = -5.71, 95% CI 2-sided [-12.43 to 1.00]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.1909, ANCOVA; Least Squares Mean Difference = -4.57, 95% CI 2-sided [-11.45 to 2.32]

20. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units per liter (U/L)
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 23 | 25 | 22
units per liter (U/L)
  ALT | -2.2 [-8.48 to 3.99] | 4.8 [-1.75 to 11.38] | 12.5 [6.30 to 18.79] | 6.6 [-0.06 to 13.32]
  AST | -1.8 [-5.50 to 1.93] | 3.2 [-0.71 to 7.12] | 6.7 [2.93 to 10.37] | 4.7 [0.77 to 8.71]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; ALT; Test type: Superiority; p = 0.1294, ANCOVA; Least Squares Mean Difference = 7.1, 95% CI 2-sided [-2.10 to 16.22]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; ALT; Test type: Superiority; p = 0.0012, ANCOVA; Least Squares Mean Difference = 14.8, 95% CI 2-sided [5.98 to 23.59]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; ALT; Test type: Superiority; p = 0.0594, ANCOVA; Least Squares Mean Difference = 8.9, 95% CI 2-sided [-0.36 to 18.11]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; AST; Test type: Superiority; p = 0.0730, ANCOVA; [Least Squares Mean Difference = 5.0, 95% CI 2-sided [-0.47 to 10.45]
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; AST; Test type: Superiority; p = 0.0020, ANCOVA; Least Squares Mean Difference = 8.4, 95% CI 2-sided [3.17 to 13.70]
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; AST; Test type: Superiority; p = 0.0200, ANCOVA; Least Squares Mean Difference = 6.5, 95% CI 2-sided [1.05 to 12.00]

21. Secondary Outcome: Change From Baseline in Leptin at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/L
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 24 | 23 | 19
μg/L | 0.95 [-1.37 to 3.27] | -0.24 [-2.66 to 2.18] | -0.57 [-2.99 to 1.85] | -3.23 [-5.90 to -0.56]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.4812, ANCOVA; Least Squares Mean Difference = -1.19, 95% CI 2-sided [-4.55 to 2.16]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.3679, ANCOVA; Least Squares Mean Difference = -1.53, 95% CI 2-sided [-4.88 to 1.83]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.0210, ANCOVA; Least Squares Mean Difference = -4.18, 95% CI 2-sided [-7.72 to -0.65]

22. Secondary Outcome: Change From Baseline in Adiponectin at the Primary Analysis Time Point
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per liter (mg/L)
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 24 | 23 | 19
milligrams per liter (mg/L) | 0.20 [-0.20 to 0.60] | 0.05 [-0.37 to 0.48] | -0.18 [-0.61 to 0.24] | -0.18 [-0.65 to 0.29]
Statistical Analysis 1: Comparison: Pooled Placebo; Test type: Superiority; p = 0.6227, ANCOVA; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.73 to 0.44]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.1950, ANCOVA; Least Squares Mean Difference = -0.38, 95% CI 2-sided [-0.97 to 0.20]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.2271, ANCOVA; Least Squares Mean Difference = -0.38, 95% CI 2-sided [-1.00 to 0.24]

23. Secondary Outcome: Change From Baseline in Subcutaneous Adipose Tissue (SAT) and Visceral Adipose Tissue (VAT) by Single Slice MRI at the Primary Analysis Timepoint
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mm^2
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 25 | 23 | 20 | 19
mm^2
  SAT | -25.61 [-156.99 to 105.76] | -8.55 [-145.57 to 128.47] | 7.31 [-139.08 to 153.70] | -41.91 [-192.12 to 108.29]
  VAT | 14.83 [-112.13 to 141.79] | 19.78 [-109.07 to 148.63] | -9.42 [-149.27 to 130.42] | 36.85 [-105.21 to 178.91]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; SAT; Test type: Superiority; p = 0.8591, ANCOVA; Least Squares Mean Difference = 17.06, 95% CI 2-sided [-173.57 to 207.69]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; SAT; Test type: Superiority; p = 0.7404, ANCOVA; Least Squares Mean Difference = 32.92, 95% CI 2-sided [-164.11 to 229.95]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; SAT; Test type: Superiority; p = 0.8711, ANCOVA; Least Squares Mean Difference = -16.30, 95% CI 2-sided [-215.50 to 182.90]
Statistical Analysis 4: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; VAT; Test type: Superiority; p = 0.9569, ANCOVA; Least Squares Mean Difference = 4.95, 95% CI 2-sided [-176.64 to 186.53]
Statistical Analysis 5: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; VAT; Test type: Superiority; p = 0.8025, ANCOVA; Least Squares Mean Difference = -24.26, 95% CI 2-sided [-216.53 to 168.02]
Statistical Analysis 6: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; VAT; Test type: Superiority; p = 0.8202, ANCOVA; Least Squares Mean Difference = 22.02, 95% CI 2-sided [-170.09 to 214.12]

24. Secondary Outcome: Change From Baseline in Waist Circumference by Single Slice MRI at the Primary Analysis Timepoint
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Groups:
- Cohort A: ISIS 703802, 20 mg Q4W: Participants received ISIS 703802, 20 mg SC once every week for 26 doses.
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg Q4W
Number analyzed (Participants) | 25 | 24 | 25 | 22
cm | -2.25 [-6.85 to 2.35] | -2.14 [-6.77 to 2.49] | -2.95 [-7.51 to 1.61] | -0.59 [-5.41 to 4.23]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.9734, ANCOVA; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-6.47 to 6.69]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.8333, ANCOVA; Least Squares Mean Difference = -0.70, 95% CI 2-sided [-7.25 to 5.86]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg Q4W; Test type: Superiority; p = 0.6207, ANCOVA; Least Squares Mean Difference = 1.66, 95% CI 2-sided [-4.99 to 8.31]

25. Secondary Outcome: Change From Baseline in Waist to Hip Ratio (WHR) at the Primary Analysis Timepoint
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 24 | 24 | 25 | 22
ratio | 0.01 [-0.03 to 0.04] | 0.01 [-0.02 to 0.05] | -0.01 [-0.04 to 0.02] | 0.01 [-0.03 to 0.05]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.8026, ANCOVA; Least Squares Mean Difference = 0.01, 95% CI 2-sided [-0.04 to 0.06]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.4917, ANCOVA; Least Squares Mean Difference = -0.02, 95% CI 2-sided [-0.07 to 0.03]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.8916, ANCOVA; Least Squares Mean Difference = 0.00, 95% CI 2-sided [-0.05 to 0.05]

26. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at the Primary Analysis Timepoint
Description: An ANCOVA model was performed on the change from Baseline to Primary Analysis Time Point.
Time Frame: Baseline, Week 27 for Cohort A, and Week 25 for Cohorts B and C
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
Number analyzed (Participants) | 26 | 24 | 25 | 22
kg/m^2 | -0.27 [-0.69 to 0.15] | -0.17 [-0.59 to 0.26] | -0.37 [-0.79 to 0.04] | -0.50 [-0.94 to -0.05]
Statistical Analysis 1: Comparison: Pooled Placebo vs Cohort B: ISIS 703802, 40 mg Q4W; Test type: Superiority; p = 0.7280, ANCOVA; Least Squares Mean Difference = 0.11, 95% CI 2-sided [-0.50 to 0.71]
Statistical Analysis 2: Comparison: Pooled Placebo vs Cohort C: ISIS 703802, 80 mg Q4W; Test type: Superiority; p = 0.7354, ANCOVA; Least Squares Mean Difference = -0.10, 95% CI 2-sided [-0.69 to 0.49]
Statistical Analysis 3: Comparison: Pooled Placebo vs Cohort A: ISIS 703802, 20 mg QW; Test type: Superiority; p = 0.4682, ANCOVA; Least Squares Mean Difference = -0.23, 95% CI 2-sided [-0.84 to 0.39]

27. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was defined as any unfavorable and unintended sign (including a clinically-significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE was considered related to the investigational drug product. TEAEs were defined as adverse events that occurred after the first administration of study drug.
Time Frame: Up to 13 weeks post treatment period (up to 39 weeks)
Population: Safety set included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A: ISIS 703802, 20 mg Q4W: Participants received ISIS 703802, 20 mg once every week for 26 doses.
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg Q4W
Number analyzed (Participants) | 27 | 26 | 26 | 26
Participants | 18 | 21 | 24 | 23

ADVERSE EVENTS:
Time Frame: Up to 13 weeks post-treatment period (up to 39 weeks)
Description: Safety population included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Pooled Placebo | Cohort B: ISIS 703802, 40 mg Q4W | Cohort C: ISIS 703802, 80 mg Q4W | Cohort A: ISIS 703802, 20 mg QW
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/27 | 1/26 | 2/26 | 1/26
Other Adverse Events (participants affected / at risk) | 13/27 | 15/26 | 20/26 | 14/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=27) | Cohort B: ISIS 703802, 40 mg Q4W (N=26) | Cohort C: ISIS 703802, 80 mg Q4W (N=26) | Cohort A: ISIS 703802, 20 mg QW (N=26)
Actinomycosis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=27) | Cohort B: ISIS 703802, 40 mg Q4W (N=26) | Cohort C: ISIS 703802, 80 mg Q4W (N=26) | Cohort A: ISIS 703802, 20 mg QW (N=26)
Injection site pruritus (General disorders) | 0 | 1 | 8 | 2
Injection site erythema (General disorders) | 0 | 1 | 6 | 2
Pyrexia (General disorders) | 0 | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 1
Urinary tract infection (Infections and infestations) | 4 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 2
Sinusitis (Infections and infestations) | 1 | 2 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 3
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 0 | 0 | 2
Vaginal infection (Infections and infestations) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2
Blood glucose increased (Investigations) | 0 | 0 | 2 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 1 | 1 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03371355/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT03371355/SAP_001.pdf